CLINICAL TRIAL: NCT01528436
Title: Umbilical Cord Blood Therapy for Cerebral Palsy: a Randomized,Double-blind, Placebo-controlled Trial
Brief Title: Umbilical Cord Blood Therapy for Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Associate Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPUCBRCT
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Umbilical Cord Blood; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umbilical Cord Blood and Rehabilitation (Experimental): Allogeneic Umbilical Cord Blood infusion and Active Rehabilitation
  Interventions: Biological: Umbilical Cord Blood Infusion; Other: Active Rehabilitation
- Placebo Umbilical Cord Blood and Rehabilitation (Active Comparator): Placebo Umbilical Cord Blood infusion and Active Rehabilitation
  Interventions: Other: Placebo Umbilical Cord Blood; Other: Active Rehabilitation

INTERVENTIONS:
Biological: Umbilical Cord Blood Infusion — The subjects will be undertaken allogeneic umbilical cord blood infusion intravenously or intraarterially under non-myeloablative immunosuppression.
  Other Names: Donated Umbilical Cord Blood Units from Affiliated Cord Blood Bank
  Arms: Umbilical Cord Blood and Rehabilitation
Other: Placebo Umbilical Cord Blood — Placebo Umbilical Cord Blood that resembles cord blood in appearance was designed.
  Arms: Placebo Umbilical Cord Blood and Rehabilitation
Other: Active Rehabilitation — All subjects should participate in active rehabilitation. They will receive two physical and occupational therapy sessions per day. Post discharge, each participant should continue to receive rehabilitation therapy at least 3 days per week until the study completion.

SUMMARY:
This randomized controlled study aims to evaluate the efficacy of umbilical cord blood therapy for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a disorder of movement and posture resulted from a non-progressive lesion or injury of the immature brain. It is a leading cause of childhood onset disability.

Many experimental animal studies have revealed that umbilical cord blood is useful to repair neurological injury in brain.

On the basis of many experimental studies, umbilical cord blood is suggested as a potential therapy for cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy with abnormal muscle tone
* Gross Motor Function Classification System (GMFCS): I, II, III, IV, V
* Willing to comply with all study procedure

Exclusion Criteria:

* Medical instability including pneumonia or renal function at enrollment
* Presence of known genetic disease
* Presence of drug hypersensitivity which is related to this study remedy
* Poor cooperation of guardian,including inactive attitude for rehabilitation and visits for follow-up
* Decision by the principal investigator when there are unexpected events including brain surgery, that may affect the outcome

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes in Motor Performance | Baseline - 1 month - 3 months
  GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, Higher value means better motor quality). We will report GMPM scores at each assessment time points.
Changes in Standardized Gross Motor Function | Baseline - 1 month - 3 months
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function). We will report GMFM scores at each assessment time points.

SECONDARY OUTCOMES:
Changes in Cognitive Neurodevelopmental Outcome | Baseline - 1 month - 3 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Mental Scales (higher value means better mental function: 0 - worst, 178 - best). We will report K-BSID-II Mental Scale raw scores at each assessment time points.
Changes in Motor Neurodevelopmental Outcome | Baseline - 1 month - 3 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Motor Scales (higher value means better motor function: 0 - worst, 112 - best). We will report K-BSID-II Motor Scale raw scores at each assessment time points.
Changes in Functional Independence in Daily Activities | Baseline - 1 month - 3 months
  WeeFIM (Functional Independence Measure for Children) measures functional independence in daily activities. WeeFIM contains 18 items and each item is ranked from complete dependence (scored as 1) to complete independence (scored as 7). The range is from 18 to 126 and higher scores mean more independent performance in daily activities. We will report total WeeFIM scores measured at each assessment time points.
Changes in Visual Perception Test | Baseline - 1 month - 3 months
  We will evaluate visual perception function with one of three measures: DTVP (Developmental Test of Visual Perception), MVPT (Motor-free Visual Perception Test), and VMI (Visual-Motor Integration, Visual Perception and Motor Coordination). All can be scored as percentile rank from 0 to 100. Higher values mean better visual perception ability.
Changes in Muscle Strength | Baseline - 1 month - 3 months
  Summation of MMT (manual muscle strength test score): summated scores of the manual muscle strength test (zero=0, trace=1, poor=2, fair=3, good=4, normal=5) for flexors, extensors, abductors, and adductors of bilateral shoulder and hip joints; flexors and extensors of bilateral elbow, wrist, and knee; dorsiflexors and plantar flexors of the ankles (range: 0 ~ 160) Higher scores mean better muscle strength. Categories of outcome table will be summation of MMT scores measured at each assessment time point.
Changes in Functional Performance in Daily Activities | Baseline - 1 month - 3 months
  Pediatric Evaluation of Disability Inventory (PEDI) for assessing functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best). We will report 2 scales and 3 domains of each scale: a Functional Skill Scale (FSS) and a Caregiver Assistance Scale (CAS) which are divided respectively into 3 domains: self care, mobility, and social function. Categories of outcome table will be each domain scores measured at each assessment time point.
Changes in Brain Glucose Metabolism Using by Brain 18F-FDG PET | Baseline - 2 weeks
  18F-FDG PET imaging will be underwent twice prior to and then 2 weeks post-treatment. All scans will be reviewed by a nuclear physician. Spatial pre-processing and statistical analyses will be done using SPM8 implanted in Matlab to compare differences in regional brain glucose metabolism between groups and differences between pre- and post-therapy imaging data. We will reported increased areas and decreased areas of glucose metabolism in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea